CLINICAL TRIAL: NCT00364572
Title: Efficacy of Epidural Etanercept in the Treatment of Sciatica
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Steve P. Cohen, Walter Reed Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WU#06-20009A
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Sciatica
Keywords: sciatica; low back pain; epidural; tumor necrosis factor
MeSH Terms: conditions — Sciatica; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Two injections of epidural saline 2 weeks apart
  Interventions: Drug: placebo (control procedure)
- Epidural injection of etanercept (Experimental): Two injections of epidural etanercept 2 weeks apart
  Interventions: Drug: epidural injection of etanercept

INTERVENTIONS:
Drug: epidural injection of etanercept — 2 injections of etanercept 2 weeks apart with doses ranging from 2 mg to 6 mg
  Arms: Epidural injection of etanercept
Drug: placebo (control procedure) — Two injections of epidural saline 2 weeks apart
  Arms: 1

SUMMARY:
Tumor necrosis factor (TNF)-alpha has been strongly implicated as a major contributing factor for the development of radiculopathy. In animal studies, the application of TNF-alpha to nerve roots results in pain behavior indicative of radiculopathy. The use of TNF-alpha inhibitors (etanercept and infliximab) have been shown to prevent this pain behavior. Open-label studies in humans have shown both etanercept and infliximab provide excellent, long-term relief in patients with acute radiculopathy from herniated disc. However, a recent placebo-controlled study failed to demonstrate any significant difference from placebo. The investigators have already established the safety of neuraxial etanercept in a trial that has just been completed (not yet published). The objective of this study is to determine whether small doses of epidural etanercept, an anti-TNF-a medication, is an effective treatment for LBP caused by nerve root irritation (i.e., radiculopathy).

DETAILED DESCRIPTION:
As per the wishes of the Dept. of the Army and Walter Reed Army Medical Center Dept. of Clinical Investigation, patients will be randomized in a 3:1 ratio to receive 2 transforaminal epidural etanercept or saline injections at 2-week intervals. Both patients and physicians will be blinded as to the injectate and treatment group. There will be 3 study groups. Group I will receive either 2 mg of etanercept or saline per injection. Group II will receive either 4 mg of etanercept or saline per injection. Group III will receive either 6 mg of etanercept or saline per injection. In each group there will be 8 patients: 6 who receive etanercept and 2 who receive saline. As per a previous study we just completed, etanercept doses will not be escalated until all 6 patients have completed their 1-month follow-up visits without any evidence of toxicity or complications.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic low back pain of radicular origin of > 2 months but < 1 year duration.
2. Failure of conservative therapy to include physical and pharmacotherapy.
3. MRI evidence of a herniated disc corresponding to the patient's radicular symptoms.
4. Normal white blood cell count (drawn in 1 blood vial).

Exclusion Criteria:

1. Uncontrolled coagulopathy.
2. Pregnancy, which will be ruled out by a urine pregnancy test if any question as to the patient's status exists.
3. Allergy to contrast dye.
4. Unstable medical condition (e.g., unstable angina or congestive heart failure).
5. Rheumatoid arthritis, Crohn's disease or spondylarthropathy.
6. Unstable neurological condition (e.g., multiple sclerosis)
7. Systemic infection
8. Age < 18 or > 70 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale pain score, Oswestry disability index, medication intake | 7 months

SECONDARY OUTCOMES:
Global perceived effect, white blood cell count | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins School of Medicine and Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Ozaktay AC, Cavanaugh JM, Asik I, DeLeo JA, Weinstein JN. Dorsal root sensitivity to interleukin-1 beta, interleukin-6 and tumor necrosis factor in rats. Eur Spine J. 2002 Oct;11(5):467-75. doi: 10.1007/s00586-002-0430-x. Epub 2002 Jun 4. PMID 12384756
- [Result] Olmarker K, Larsson K. Tumor necrosis factor alpha and nucleus-pulposus-induced nerve root injury. Spine (Phila Pa 1976). 1998 Dec 1;23(23):2538-44. doi: 10.1097/00007632-199812010-00008. PMID 9854752
- [Result] Olmarker K, Nutu M, Storkson R. Changes in spontaneous behavior in rats exposed to experimental disc herniation are blocked by selective TNF-alpha inhibition. Spine (Phila Pa 1976). 2003 Aug 1;28(15):1635-41; discussion 1642. doi: 10.1097/01.BRS.0000083162.35476.FF. PMID 12897484
- [Result] Igarashi T, Kikuchi S, Shubayev V, Myers RR. 2000 Volvo Award winner in basic science studies: Exogenous tumor necrosis factor-alpha mimics nucleus pulposus-induced neuropathology. Molecular, histologic, and behavioral comparisons in rats. Spine (Phila Pa 1976). 2000 Dec 1;25(23):2975-80. doi: 10.1097/00007632-200012010-00003. PMID 11145807
- [Result] Korhonen T, Karppinen J, Malmivaara A, Autio R, Niinimaki J, Paimela L, Kyllonen E, Lindgren KA, Tervonen O, Seitsalo S, Hurri H. Efficacy of infliximab for disc herniation-induced sciatica: one-year follow-up. Spine (Phila Pa 1976). 2004 Oct 1;29(19):2115-9. doi: 10.1097/01.brs.0000141179.58778.6c. PMID 15454701
- [Result] Korhonen T, Karppinen J, Paimela L, Malmivaara A, Lindgren KA, Jarvinen S, Niinimaki J, Veeger N, Seitsalo S, Hurri H. The treatment of disc herniation-induced sciatica with infliximab: results of a randomized, controlled, 3-month follow-up study. Spine (Phila Pa 1976). 2005 Dec 15;30(24):2724-8. doi: 10.1097/01.brs.0000190815.13764.64. PMID 16371894
- [Result] Genevay S, Stingelin S, Gabay C. Efficacy of etanercept in the treatment of acute, severe sciatica: a pilot study. Ann Rheum Dis. 2004 Sep;63(9):1120-3. doi: 10.1136/ard.2003.016451. Epub 2004 Apr 28. PMID 15115710
- [Result] Cohen SP, Griffith S, Larkin TM, Villena F, Larkin R. Presentation, diagnoses, mechanisms of injury, and treatment of soldiers injured in Operation Iraqi Freedom: an epidemiological study conducted at two military pain management centers. Anesth Analg. 2005 Oct;101(4):1098-1103. doi: 10.1213/01.ane.0000169332.45209.cf. PMID 16192528
- [Derived] Cohen SP, Bogduk N, Dragovich A, Buckenmaier CC 3rd, Griffith S, Kurihara C, Raymond J, Richter PJ, Williams N, Yaksh TL. Randomized, double-blind, placebo-controlled, dose-response, and preclinical safety study of transforaminal epidural etanercept for the treatment of sciatica. Anesthesiology. 2009 May;110(5):1116-26. doi: 10.1097/ALN.0b013e3181a05aa0. PMID 19387178